CLINICAL TRIAL: NCT06556472
Title: Safety and Efficacy of Continuous Infusion of Terlipressin With Norepinephrine Versus Norepinephrine Alone in Improving Outcomes of Acute Kidney Injury in Acute on Chronic Liver Failure With Septic Shock - A Randomised Controlled Trial
Brief Title: Safety and Efficacy of Continuous Infusion of Terlipressin With Norepinephrine Versus Norepinephrine Alone in Improving Outcomes of Acute Kidney Injury in Acute on Chronic Liver Failure With Septic Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-19
Record Dates: First submitted 2024-07-30; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Terlipressin; Nordefrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous terlipressin infusion + Norepinephrine (Experimental): 1. Patients in this group will receive continuous terlipressin infusion (1 mg/24 hr on day 1, increasing to 1 mg in 24 hours if target MAP not achieved ,reaching maximum terlipressin dose of 4 mg/24 hr on day 4).If target MAP not achieved by terlipressin dose ,increase noradrenaline dose keeping terlipressin maximum 1 mg ,2 mg ,3mg ,4mg at Day 1,2,3,4 respectively.
  2. Norepinephrine will be initiated @0.05mcg/kg/min and titrated upto 0.5 mcg/kg/min to maintain a MAP > 65 to 75 mm Hg.
  3. IV albumin as per volume status to maintain target MAP .
  4. If the target MAP is not achieved, a third vasopressor along with hydrocortisone, Adrenaline and then phenylephrine.
  Interventions: Drug: Terlipressin; Drug: Norephrine
- Norepinephrine (Active Comparator): 1. Patients in this group will receive norepinephrine only, with a dose range of 0.05 mcg/kg/min to 0.5 mcg/kg/min to maintain a MAP > 65 to 75 mm Hg.
  2. IV albumin as per volume status to maintain target MAP .
  3. If the target MAP is not achieved, vasopressin along with hydrocortisone, followed by adrenaline and phenylephrine, may be added as a fourth vasopressor.
  Interventions: Drug: Norephrine

INTERVENTIONS:
Drug: Terlipressin — 1. Patients in this group will receive continuous terlipressin infusion (1 mg/24 hr on day 1, increasing to 1 mg in 24 hours if target MAP not achieved ,reaching maximum terlipressin dose of 4 mg/24 hr on day 4).If target MAP not achieved by terlipressin dose ,increase noradrenaline dose keeping terlipressin maximum 1 mg ,2 mg ,3mg ,4mg at Day 1,2,3,4 respectively.
  Arms: Continuous terlipressin infusion + Norepinephrine
Drug: Norephrine — 1. Patients in this group will receive norepinephrine only, with a dose range of 0.05 mcg/kg/min to 0.5 mcg/kg/min to maintain a MAP > 65 to 75 mm Hg.

SUMMARY:
ACLF is defined differently in APASL,EASL and AASLD.APASL talks of reversibility in ACLF as per its definition and constitution of Homogenous population with ACLF.The definition of ACLF as per APASL is an acute hepatic insult manifesting as jaundice (serum bilirubin ≥ 5 mg/dL (85 micromol/L) and coagulopathy (INR ≥ 1.5 or prothrombin activity < 40%) complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease/cirrhosis, and is associated with a high 28-day mortality.

At the onset of septic shock there is initially an increased secretion of Arginine vasopressin. However, this initial rise is short lasting, and the vasopressin levels come back to normal or low serum levels with continued hypotension. However, even normal levels are too low for the degree of hypotension in septic shock. This causes a relative deficiency of vasopressin in septic shock. The exact time when this fall happens is not known and it is likely to be variable. Vasopressin was therefore tried as an agent in septic shock. Terlipressin is a synthetic analogue of vasopressin. It has a greater selectivity for the V1 receptor.

Currently, Norepinephrine is recommended as the first vasopressor to be started in general in septic shock population.(3) Catecholamines are the clinically used vasopressor agents of choice for supporting arterial blood pressure and ensuring adequate organ perfusion.

Development of adrenergic hyposensitivity with loss of catecholamine presser effects is seen in advanced stages of Vasodilatory Shock. Progressively increasing catecholamine therapy frequently enters into a vicious cycle of major adverse side effects resulting in continuous clinical deterioration necessitating further catecholamine excess.

DETAILED DESCRIPTION:
• Aim: To study the safety and efficacy of low-dose continuous infusion of terlipressin with norepinephrine compared to norepinephrine alone in improving outcomes of Acute kidney injury occurring in the context of septic shock in patients with Acute on chronic liver failure.

Study population:

1. septic shock with AKI in patients of ACLF

   Study design: Prospective open labelled randomised controlled study. The study will be conducted in Department of Hepatology ILBS- intensive care unit.

   At admission:

   Complete history and physical examination

   - Recent Diuretics use

   - Loose stools / Recurrent vomiting
   * Fever, signs of sepsis (Systemic inflammatory response syndrome), shock, respiratory tract infection,spontaneous bacterial peritonitis
   * Recent contrast use (< 7 days)/ nephrotoxins use including NSAIDs
   * Prior renal dysfunction, chronic kudney disease, history of Hemodialysis
   * History of Hypertension, Diabetes/ renal stones
   * Baseline workup for Acute on chronic liver failure
   * Severity of liver disease,AARC-ACLF, MELD score, CTP score (B) Intervention during 0-3 hours (Before randomization) - Pre-randomization interventions:
   * Withdrawal of diuretics/ Withdrawal of lactulose (in patients with loose stools)
   * IV hydration with 5 % albumin according to FRISC protocol
   * Urine output monitoring (catheterize and monitor hourly) ,hourly MAP, Pulse rate
   * Use of broad-spectrum IV antibiotics promptly within the first hour, in case of suspected/proven sepsis (Avoid nephrotoxic drugs as possible)
   * Lung ultrasound and IVC (Inferior Vena Cava) measurements will be performed at baseline and hourly for 3 hours.
   * Fluid boluses will be administered based on IVC measurements and lung ultrasound findings.
   * Fluid bolus criteria include IVCCI(inferior vena cava collapsibility index) >40% and an A profile on lung ultrasound.
   * The stopping rule for fluid boluses is IVCCI <40% or a B profile on lung ultrasound.
   * Patients showing improvement within 3 hours will be excluded from further intervention

   Monitoring • Hemodynamic- MAP,HR, Urine output hourly

   • Metabolic - lactate, blood sugar, electrolytes

   • Microbiologic - urine -routine, microscopy and culture, ascitic fluid analysis along with gram stain and c/s in blood culture bottle, sputum or mini BAL -C/s Gram stain. Daily.

   • Others - daily chest X-ray, Procalcitonin, Cardiac-ECG, 2D echo. Prognostic models: CTP, MELD SOFA daily

   Stopping Rule

   • Requirement of Third Vasopressor (Need of Norepinephrine > 0.5 mcg/kg/min):

   • If a patient requires norepinephrine at a dose exceeding 0.5 mcg/min, indicating the need for a third vasopressor, this criterion triggers specific actions as per the study protocol.

   • Threshold (Stopping Rule) for Fluid Boluses:

   • Fluid boluses will be administered based on IVC and lung ultrasound findings.

   • The stopping rule for fluid boluses is activated if any of the following criteria are met:

   • IVC >25

   • IVCCI <40%

   • B profile on lung ultrasound

   • Severe Side Effects or Toxicities (CTAE Grade 4):

   • If a patient experiences severe side effects or toxicities categorized as CTAE (Common Terminology Criteria for Adverse Events) Grade 4, including arrhythmia, AMI (Acute Myocardial Infarction), cardiomyopathy (as defined later), cyanosis, suspicion or confirmed bowel ischemia, or any other severe adverse event, specific actions or interventions may be required.

   Salvage group • Patient Unwilling for Further Hospital Stay: • Non responders or when patient in either arm failed

   • Study will be stopped and management will be done accordingly to guidelines

   • Adverse effects to terlipressin
   * Further increase in MAP to be maintained by addition of other ( vasopressors--vasopressin, phenylephrine,steroids)
   * If the target MAP is not achieved in arm A ,a third vasopressor along with hydrocortisone, Adrenaline and then phenylephrine
   * If the target MAP is not achieved in arm B, vasopressin along with hydrocortisone, followed by adrenaline and phenylephrine, may be added as a fourth vasopressor.
   * The indication for start of steroid
   * Maximum dose of vasopressor in each arm and all patients in salvage arm
   * Hydrocortisone 100-150mg bolus start followed by 50mg q6hrly and later tapering dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years and <60 yrs
2. ACLF as per APASL
3. AKI according to KDIGO Criteria
4. septic shock requiring norepinephrine (<0.05mcg/kg/min).

Exclusion Criteria:

1. Septic shock requiring 2 vasopressors (Norephinephrine reuirement > 0.05mcg/kg/min)
2. Symptomatic cardiopulmonary disease
3. Chronic kidney disease
4. Peripheral vascular disease
5. Hepatocellular carcinoma outside Milan criteria
6. Prior use of terlipressin in last 48 hours
7. Patients with hypovolemic or hemorrhagic shock
8. Patients already meeting criteria for dialysis or with history of dialysis in last 7 days
9. Intrinsic kidney disease, Acute tubular necrosis with urinary output < 400 ml /day or obstructive uropathy
10. History of immunosuppressive drugs
11. Pregnancy
12. Human immunodeficiency virus 1 and 2
13. Portal vein thrombus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing 1 stage improvement in Acute kidney injury stage with resolution of shock at day 4 in both groups | Day 4

SECONDARY OUTCOMES:
Outcome of acute kidney injury at day 4,7 | Day 4 and 7
  Outcome in terms of resolution, persistence or progreession
Incidence of adverse events in both groups | 1 year
Need of renal replacement therapy at day 7 | Day 7
Duration of ICU and hospital stay | 1 year
Mortality | Day 7 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided